CLINICAL TRIAL: NCT02036034
Title: Effectiveness of Modified Ophthalmic Draping Method in Preventing Carbon Dioxide Accumulation in Patient Undergoing Eye Surgery Under Local Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Alvin Tan Siaw Boon, Lecturer, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: eyedrapCO2
Record Dates: First submitted 2011-08-15; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2011-08

CONDITIONS: To Prevent Hypercarbia Under the Opthalmology Drape During Surgery.; To Prevent Hypothermia During Opthalmology Surgery.

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drape with forced air warmer (Active Comparator): forced air warmer placed under the chin before draping, inflated after draping completed.
  Interventions: Device: forced air warmer (Bair Hugger)
- drape with warming blanket (Placebo Comparator): warming blanket placed on torso of patient under the drape.
  Interventions: Device: warming blanket

INTERVENTIONS:
Device: forced air warmer (Bair Hugger) — forced air warmer placed under the chin before draping, forced air warmer inflated after draping is completed.
  Other Names: Forced air warmer brand - Bair Hugger
  Arms: drape with forced air warmer
Device: warming blanket — warming blanket placed on torso of patient under the drape.
  Other Names: warming blanket brand - Thermamed warming system
  Arms: drape with warming blanket

SUMMARY:
The investigators hypothesize that this modified ophthalmic draping will reduce the accumulation and rebreathing of carbon dioxide during eye surgery.

DETAILED DESCRIPTION:
Majority of eye surgery has been widely done under local anesthesia provided by the ophthalmologist with or without sedation.The surgical drapes used often covers the patients face and beyond in order to maintain sterility of the surgical field. This can lead to accumulation of carbon dioxide under ophthalmic drapes due to the exhaled carbon dioxide escapes incompletely through the drapes;hence results in an increase of carbon dioxide in the ambient air surrounding the patient's head.This causes an increase in arterial carbon dioxide partial pressure and thus hyperventilation and patient discomfort with restlessness and unable to stay still during the surgery.

In recent years,several types of ophthalmic drapes have been produced.This study is look for possible difference in accumulation of carbon dioxide under the standard ophthalmic drapes compared to the modified draping.

ELIGIBILITY:
Inclusion Criteria:

- ASA physical status I,II OR III,adult aged 40 to 80 years old,scheduled to undergo elective eye surgery under local anaesthetic at UMMC will be enrolled in this study.

Exclusion Criteria:

* Pre-existing pulmonary disease,psychological disorders,neurological disorder and patient required sedation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
transcutaneous CO2 level in mmHg under surgical drape with forced air warmer | 10 minutes, 15 minutes, 30 minutes
  baseline transcutanoeus CO2 level will be taken before surgical draping. After draping, CO2 level will be measured with transcutaneous CO2 frome earlobe at 10 minutes, 15 minutes, and 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Siaw Boon Tan, Principal Investigator — Universiti Malaya; sukhcharanjit S Singh, Study Chair — Universiti Malaya
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia